CLINICAL TRIAL: NCT03549533
Title: Impact of Aluminum on Sperm DeoxyriboNucleic Acid (DNA) Quality
Brief Title: Impact of Aluminum on Sperm DNA Quality
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1708031; 2017-A01825-48 (Other: ANSM)
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Insemination, Artificial
Keywords: Aluminum; Sperm; DNA methylation; DNA fragmentation; Seminal plasma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Samples of sperm will be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- artificial insemination: Patient who perform his first artificial insemination will be included. Samples of sperm will be analyzed.
  Interventions: Other: samples of sperm

INTERVENTIONS:
Other: samples of sperm — As in the usual practice during artificial insemination a samples of sperm will be collected and analyzed.

SUMMARY:
Between 1950 and 2013, aluminum production was multiplied by thirty in the world. Today, men's exposure to aluminum, including food products, cosmetics, air and water contamination, and a number of drugs (vaccine, gastric bandages, etc.) has never been so high and should continue to increase. At the same time, we are witnessing a decline in male fertility in Western countries.

In this context, several teams, including ours, have studied the impact of aluminum on the fertility of men. These studies have shown that aluminum accumulates in semen and especially in sperm near its DNA.

Aluminum has already shown that it is capable of damaging the DNA of various cells, especially to increase DNA fragmentation. We therefore hypothesize that aluminum could lead to increased sperm DNA fragmentation. This would result in a decrease of men fertility and in higher risk of miscarriage.

DETAILED DESCRIPTION:
In order to confirm this hypothesis, this study aims to dose aluminum in the spermatozoa of 80 patients who perform artificial insemination and correlate this result to their sperm DNA fragmentation. Patients will be recruited from the reproductive biology unit of Saint-Etienne University Hospital. Aluminum assays will be carried out using an Atomic Absorption Spectrophotometry technique by Prof. Exley at Keele University in Great Britain, a world expert in aluminum toxicity. Measurements of sperm DNA damage will be carried out using flow cytometry by our research team (SAINBIOSE INSERM U1059) at the Medecine Faculty of Saint-Etienne.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to a social security scheme
* Patient who perform his first artificial insemination
* Patient who is 18 years old or more

Exclusion Criteria:

* Patient having expressed his refusal to participate in the study after information on the protocol and delivery of an information notice.
* Patient for whom the total quantity of spermatozoa is not sufficient for separation by ascending migration (in this case all the spermatozoa from the pellet are used for the insemination)
* Patient under justice protection (guardianship)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who perform his first artificial insemination
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Aluminum content of sperm | Day 1
  To analyze concentration of aluminum content of sperm the day of inclusion. Aluminum content of sperm will be measured by atomic absorption spectrophotometry.
Spermatic DNA fragmentation | Day 1
  To analyze Spermatic DNA fragmentation. Spermatic DNA fragmentation will be measured by flow cytometry technical.

SECONDARY OUTCOMES:
Spermatic DNA methylation | Day 1
  To analyze Spermatic DNA fragmentation. Spermatic DNA fragmentation will be measured by flow cytometry technical.
Aluminum content of seminal plasma | Day 1
  To analyze aluminum content of seminal plasma. Aluminum content of seminal plasma will be measured by atomic absorption spectrophotometry.
HCG value | Weeks 2
  To analyze HCG value in the patient women. HCG value will be measured by blood sample two weeks after artificial insemination
Spontaneous Miscarriage | Months 9
  Analyze the rate of spontaneous miscarriage.
Live birth | Months 9
  Analyze the rate of live birth

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe KLEIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No